CLINICAL TRIAL: NCT03397654
Title: A Phase Ib Study of Pembrolizumab Following Trans-Arterial Chemoembolization in Primary Liver Carcinoma
Brief Title: Study of Pembrolizumab Following TACE in Primary Liver Carcinoma
Acronym: PETAL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PETAL1
Record Dates: First submitted 2017-12-01; First posted 2018-01-12 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Primary Liver Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TACE followed by pembrolizumab (Experimental): Trans-arterial chemoembolization (TACE) using doxorubicin solution (60 mg dose) and gelatin sponge particles; followed, at least 30 or 45 days later, by pembrolizumab solution (200 mg dose) every 3 weeks for a maximum of 1 year
  Interventions: Drug: Pembrolizumab; Combination Product: Trans-arterial chemoembolization

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab solution
  Other Names: KEYTRUDA
Combination Product: Trans-arterial chemoembolization — Doxorubicin injected through the hepatic blood supply directly to the cancer-affected part of the liver, then gelatin sponge particles injected to block the blood vessels supplying the tumour
  Other Names: TACE

SUMMARY:
Open label, single arm, multi-centre study of pembrolizumab following trans-arterial chemoembolization (TACE). Twenty-six to 32 evaluable participants with primary liver cancer (hepatocellular cancer; HCC) will be assessed. The primary objective is to determine the safety and tolerability of pembrolizumab following TACE. The secondary objective is to evaluate the efficacy of pembrolizumab following TACE by improving progression-free survival rates as measured by modified response evaluation criteria in solid tumours (mRECIST) criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Be willing to provide tissue from an excisional biopsy of a tumour lesion.
4. Have at least one uni-dimensional lesion measurable by Computed Tomography (CT)-scan or Magnetic Resonance Imaging (MRI) based on mRECIST criteria.
5. Be ineligible for surgical resection or liver transplantation.
6. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
7. Demonstrate adequate organ function
8. Have an overall Child-Pugh score <7
9. Female subject of childbearing potential should have a negative urine or serum pregnancy. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Women of childbearing potential must be willing to use a highly effective method of contraception as outlined in Section 6.9.2 for the course of the study through 120 days after the last dose of Investigational Medicinal Product (IMP). Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Sexually active males must agree to use an adequate method of contraception as outlined in Section 6.9.2 starting with the first dose of IMP through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Has extrahepatic metastasis.
2. Prior TACE or systemic anticancer treatment for HCC.
3. Has any contraindication for TACE including portosystemic shunt, hepatofugal blood flow, known severe atheromatosis.
4. Has history of bleeding within the 4 weeks preceding study enrolment.
5. Has hepatic encephalopathy.
6. Has ascites that is refractory to diuretic therapy.
7. Has documented occlusion of the hepatic artery or the main portal vein (segmental portal vein thrombosis does not represent exclusion criterion provided this does not contraindicate TACE).
8. Is currently participating and receiving therapy or has participated or is participating in a study of an IMP or used an investigational device within 4 weeks of the first dose of IMP.
9. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy.
10. Has a known history of active Bacillus Tuberculosis (TB)
11. Hypersensitivity to Pembrolizumab or any of its excipients.
12. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Has known history of, or any evidence of active, non-infectious pneumonitis.
15. Has an active infection requiring systemic therapy. Exceptions relating to Hepatitis B and C virus infection are documented in Section 5.3.1, Table 5.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Principal Investigator (PI).
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through to 120 days after the last dose of IMP.
19. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PDL2 agent.
20. Has a known history of Human Immunodeficiency Virus (HIV; HIV 1/2 antibodies).
21. Has received a live vaccine within 30 days of first dose of IMP administration. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fessas P, Scheiner B, D'Alessio A, M Fulgenzi CA, Korolewicz J, Ward C, Tait P, Thomas R, Cortellini A, Sharma R, Pinato DJ. PETAL protocol: a phase Ib study of pembrolizumab after transarterial chemoembolization in hepatocellular carcinoma. Future Oncol. 2023 Mar;19(7):499-507. doi: 10.2217/fon-2022-0916. Epub 2023 Apr 25. PMID 37097715

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TACE Followed by Pembrolizumab
Started | 26
Completed | 15
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | TACE Followed by Pembrolizumab
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: Years] | 72 [63.5 to 75.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15
Eastern Cooperative Oncology Group performance [Count of Participants; unit: Participants] — Unit of measure for ECOG is 0-5
  Grade Description 0 Normal activity. Fully active
  1. Restricted in physically strenuous activity, but able to carry out work of a light or sedentary nature
  2. In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities.
  3. In bed >50% of the time. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. 100% bedridden. Completely disabled. Totally confined to bed or chair.
  5. Dead
  Participants
    ECOG 0 | 9
    ECOG 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (Safety and Tolerability)
Description: The safety and tolerability of pembrolizumab will be assessed by recording the incidence of adverse events (AEs) using National Cancer Institute Common Terminology Criteria for Adverse Events version 4 (NCI CTCAE v4).
Time Frame: from the first pembrolizumab administration to up to 130 days after the last dose, 1.5 years
Population: Patients with liver confirmed Hepatocellular carcinoma
Measure: Count of Participants; unit: Participants
Arm/Group | TACE Followed by Pembrolizumab
Number analyzed (Participants) | 15
Participants | 15

2. Secondary Outcome: Progression-free Survival Rate (PFS; Efficacy) at 12 Weeks
Description: PFS was defined by the time from last TACE to the first occurrence of documented disease progression based on RECIST v1.1 criteria or death from any cause, whichever occurred first, and it was calculated using Kaplan-Meier.
Time Frame: 12 weeks
Population: Patients with liver confirmed Hepatocellular carcinoma
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | TACE Followed by Pembrolizumab
Number analyzed (Participants) | 15
Percentage | 93.3 [82 to 100]

ADVERSE EVENTS:
Time Frame: Through study completion , an average of 1.5 years.
Description: CTCAE version v5
Arm/Group | TACE Followed by Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 10/15
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TACE Followed by Pembrolizumab (N=15)
Fatigue (General disorders) | 1
Anorexia (General disorders) | 1
Skin rash (Skin and subcutaneous tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Flu-like symptoms (General disorders) | 1
Bilirubin increase (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TACE Followed by Pembrolizumab (N=15)
Fatigue (General disorders) | 10
Anorexia (General disorders) | 10
Skin rash (Skin and subcutaneous tissue disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Lethargy (General disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 5
Peripheral oedema (Skin and subcutaneous tissue disorders) | 5
Peripheral neuropathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Flu-like symptoms (General disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Bilirubin increase (Gastrointestinal disorders) | 3
Mucositis (Gastrointestinal disorders) | 3
Dysgeusia (Gastrointestinal disorders) | 3
Hypothyroidism (Gastrointestinal disorders) | 3
Hypothyroidism (Endocrine disorders) | 3
Upper respiratory infection (Infections and infestations) | 3

LIMITATIONS AND CAVEATS:
Limitations include, limited sample size, lack of control arm and the Impact of Coronavirus disease pandemic, which made recruitment and retention of participants to the investigator-led clinical trial difficult, leading to reduction in the number of sample available for translational analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT03397654/Prot_SAP_001.pdf